CLINICAL TRIAL: NCT06344117
Title: Assessment of Volatile Organic Compounds (VOC) for the Diagnosis of Invasive Aspergillosis (IA) in Lung Transplant Recipients A Prospective Pilot Study
Brief Title: Assessment of Volatile Organic Compounds (VOC) for the Diagnosis of Invasive Aspergillosis (IA) in Lung Transplant Recipients
Acronym: UHN
Status: Recruiting | Type: Observational
Sponsor: Owlstone Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: MF3 UHN (IA)
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Invasive Aspergillosis
Keywords: Invasive Aspergillosis; VOC; Breath; Lung Transplant

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Respiratory droplets
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Controls: patients without evidence of Aspergillus colonization or Aspergillus related disease
- Colonised Aspergillus: patients with Aspergillus colonization
- Invasive Aspergillus: patients with proven or probably IA

SUMMARY:
Prospective observational pilot study to evaluate the utility of breath VOCs to detect invasive aspergillosis in lung transplant recipients that are suspected of invasive fungal disease (IFD).

DETAILED DESCRIPTION:
Invasive aspergillosis (IA) remains a major cause of morbidity and mortality in immunosuppressed patients. The diagnosis of IA is challenging due to lack of sensitive and specific clinical and radiological signs, and tissue biopsy is often precluded in many patients. Culture and microscopy of respiratory tract samples are relatively insensitive diagnostic tests. Early detection of IA can lead to specific therapeutic strategies and improved patient outcomes. Breath is a rich and complex sampling medium containing both volatile organic compounds (VOCs) and respiratory droplets carrying non-volatiles, proteins, lipids, viruses and even bacteria. The major advantage of exhaled breath analysis is non-invasiveness, with existing sampling methods already readily available.

The diagnostic or prognostic value of exhaled breath analysis has been evaluated in many respiratory diseases, including asthma, Chronic Obstructive Pulmonary Disease, idiopathic pulmonary fibrosis, as well as in some lung infections such as bacterial pneumonia. In the particular field of aspergillosis diagnosis, using a chromatographic-mass spectrometry analysis of exhaled breath in immunocompromised hosts (organ transplantation, hematological malignancies or HSCT), researchers have been able to identify an exhaled breath metabolic signature (made of β-trans-bergamotene, α-trans-bergamotene, a β-vatirenene-like sesquiterpene, and trans-geranylacetone) that potentially allows the discrimination of probable or proven aspergillosis from other lung infections, with high levels of sensitivity and specificity. Exhaled breath therefore appears as a promising field for the improvement of IA diagnosis, and more broadly of respiratory infections. Volatile organic compound (VOC) detection via thermal desorption/gas chromatography-mass spectrometry has emerged as a promising tool for early diagnosis of IA, however the sample sizes have been limited. As such, the proposed pilot study aims to identify potential VOC biomarkers for both IA and Aspergillus colonization and assess the feasibility of VOCs on breath for the diagnosis of IA in lung transplant recipients.

ELIGIBILITY:
Inclusion Criteria: Patients with the following criteria will be included in the study:

1. Over the age of 18 years
2. Recipient of single/double lung transplant
3. Willingness to participate in the study
4. Suspected of invasive fungal disease or undergo surveillance appointments
5. Capable of providing sample
6. Capable of providing consent

   -

Exclusion Criteria: Patients with the following criteria will be excluded from the study:

1. On mechanical ventilation, oxygen supplementation including nasal cannula; simple, fixed, or non-rebreathing face mask at presentation.
2. Admitted to the intensive care unit at presentation.
3. The subject is currently diagnosed with a confirmed bacterial or viral respiratory infection or has received a diagnosis of a respiratory viral or bacterial infection within the last 4 weeks.
4. Previous diagnosis of Cystic Fibrosis
5. Use of antifungals in previous 4 weeks
6. Has been previously diagnosed with respiratory fungal infection other than aspergillus within the last 3 months upon presentation.
7. Declines participation in the study.
8. On mold antifungal for >72 hours.

   -

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Lung transplant recipient patients undergoing bronchoscopy as a standard of care for suspected invasive fungal disease (IFD) or surveillance appointments will be eligible for screening.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Identifying a statistical relationship between Volatile Organic Compounds detection and the diagnosis of IA by existing International Society for Heart and Lung Transplantation (ISHLT) and MSG/EORTC criteria. | 18 months
  Identifying a statistical relationship between Volatile Organic Compounds detection and the diagnosis of IA by existing International Society for Heart and Lung Transplantation (ISHLT) and European Organization for Research and Treatment of Cancer/Mycoses Study Group (MSG/EORTC) criteria.

SECONDARY OUTCOMES:
Identifying a statistical relationship between the set of VOCs found in exhaled breath and the diagnosis of Aspergillus colonization as defined by ISHLT criteria | 18 months
  Identifying a statistical relationship between the set of VOCs found in exhaled breath and the diagnosis of Aspergillus colonization as defined by ISHLT criteria

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Husain, MD,MS, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided